CLINICAL TRIAL: NCT06134232
Title: An Open -Label, Multicenter Study of Subjects With Metastatic Castrate-Resistant Prostate Cancer Treated With PROVENGE ® and Boosted With A Single Infusion of Sipuleucel-T to Measure Immune Response
Brief Title: Metastatic Castrate-Resistant Prostate Cancer Subjects Treated With PROVENGE® + One Infusion of Sipuleucel-T
Acronym: ProvONE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dendreon (Industry)
Collaborators: WCG IRB (Unknown); Talosix (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P23-1
Record Dates: First submitted 2023-10-18; First posted 2023-11-18 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Keywords: Single Dose; Sipuleucel-T; Immune Response Rate; Safety; Adenocarcinoma of the Prostate
MeSH Terms: interventions — sipuleucel-T

STUDY DESIGN:
Intervention Model Description: AN OPEN-LABEL, MULTICENTER STUDY OF SUBJECTS WITH METASTATIC CASTRATE-RESISTANT PROSTATE CANCER TREATED WITH PROVENGE AND BOOSTED WITH A SINGLE INFUSION OF SIPULEUCEL-T TO MEASURE IMMUNE RESPONSE
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Booster Arm (Experimental): Experimental: Treatment Group: Single Infusion of Sipuleucel-T (Booster) Sipuleucel-T is an autologous cellular immunotherapy available as a suspension for intravenous infusion.
  Subjects randomized to sipuleucel-T arm will receive 1 infusion of sipuleucel-T 6-9 months after receiving commercial Provenge. These subjects will be followed as described in the schedule of events.
  Interventions: Drug: Sipuleucel-T Injection
- No Booster (No Intervention): No Intervention: Control Arm Subjects randomized to the control arm after receiving commercial Provenge will be followed as described in the schedule of events.

INTERVENTIONS:
Drug: Sipuleucel-T Injection — Single Infusion
  Arms: Booster Arm

SUMMARY:
A multicenter, open-label, prospective study to investigate immune boost response changes in patients with metastatic castrate-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
Those enrolled in the Booster Study will have had their course of treatment with PROVENGE® immunotherapy and then randomized to the Booster Study to be treated with a single booster dose of sipuleucel-T.

ELIGIBILITY:
Inclusion Criteria:

For a subject to be eligible for participation in this study, all of the following criteria must be satisfied:

1. Potential subjects are men aged ≥18 years who are clinically indicated for treatment with PROVENGE® (asymptomatic or minimally symptomatic metastatic castrate-resistant [hormone refractory] prostate cancer).
2. Have qualified for on-label PROVENGE® infusion
3. Have received all 3 infusions of PROVENGE® prior to randomization
4. Written informed consent provided prior to the initiation of study procedures
5. Estimated life expectancy ≥12 months

Exclusion Criteria:

A subject will not be eligible for participation in this study if any of the following criteria apply.

1. Men who are not clinically indicated for treatment with PROVENGE® (asymptomatic or minimally symptomatic metastatic castrate-resistant [hormone refractory] prostate cancer).
2. Need for systemic chronic immunosuppressive therapy, including antitumor necrosis factor alpha monoclonal antibodies, glucocorticoids, systemic steroids, blood products, GM-CSF or granulocyte colony-stimulating factor (G-CSF), any vaccinations, or experimental and investigational therapies (see Section 6.3.1)
3. Uncontrolled, concurrent illness, including, but not limited to the following: ongoing or active infection (bacterial, viral, or fungal), or psychiatric illness that would limit compliance with study requirements, as well as any condition that would preclude a subject from completing PROVENGE® or sipuleucel-T treatment.
4. On experimental or investigational therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male at birth
Enrollment: 400 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Assess humoral immune response to PAP and PA2024 after booster infusion | Once all subjects have completed the study through the 5 year Overall Survival Period
  To assess the humoral response ((i.e. antibody titer) to PAP and PA2024 after booster infusion in subjects with metastatic castrate-resistant prostate cancer who have received a single booster dose of sipuleucel-T vs those subjects who have not

SECONDARY OUTCOMES:
Evaluate the incidence of adverse events including laboratory abnormalities after a single booster does of sipuleucel-T | Once all subjects have completed the study through the 5 year Overall Survival Period
  For all subjects enrolled in the study. Evaluation will include descriptive statistics by treatment arm and in the aggregate of the incidence of adverse events (Number of participants with adverse events (AEs), and the incidence of clinically significant laboratory abnormalities (Number of participants experiencing clinically significant laboratory abnormalities) after initial treatment and booster (Week 28) within and between groups.
Evaluate Overall Survival | Once all subjects have completed the study through the 5 year Overall Survival Period. To evaluate safety by determining the incidence of adverse events (AEs), assessing laboratory data for clinically significant laboratory abnormalities, and evaluating
  Overall survival after booster infusion of sipuleucel-T defined as the time from randomization to death due to any cause.

OTHER OUTCOMES:
Assess biomarkers of response to treatment | Once all subjects have completed the study through the 5 year Overall Survival Period
  Biomarkers, such as cytokines, will be assessed for response to booster treatment using appropriate descriptive statistics assessed over time and at Week 28. Nominal p-values will be provided without multiplicity adjustment .appropriate descriptive statistics assessed over time and at Week 28.
Assess Antigen Response | Once all subjects have completed the study through the 5 year Overall Survival Period
  Comparison of (over time and at Week 38), the number of subjects per treatment arm with PAP and PA2024 antigen positive response using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Sheikh, PhD, Study Director — Dendreon Pharmaceuticals, LLC; Benjamin Lowentritt, MD, Study Chair — Chesapeake Urology
Locations (31):
- United States (31):
  - Arizona Urology Specialists, Tuscon, Arizona
  - City of Hope - National Medical Center, Duarte, California
  - Urology Associates of Central California Medical Group, Fresno, California
  - Unio Health Partners - Genesis Research, LLC, San Diego, California
  - Colorado Urology, Lakewood, Colorado
  - Advanced Urology Institute, Daytona Beach, Florida
  - Advanced Urology Institute, Largo, Florida
  - Advanced Urology Institute, Ocala, Florida
  - Florida Urology Partners, Riverview, Florida
  - Associated Urological Specialists, Chicago Ridge, Illinois
  - UroPartners, Glenview, Illinois
  - Advanced Urology Associates, New Lenox, Illinois
  - Urology of Indiana, Carmel, Indiana
  - First Urology, Jeffersonville, Indiana
  - Urologic Specialists of Northwest Indiana, Merrillville, Indiana
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Michigan Institute of Urology, Troy, Michigan
  - Specialty Clinical Research of St. Louis, St Louis, Missouri
  - Integrated Medical Professionals, North Hills, New York
  - Associated Medical Professionals of NY, Syracuse, New York
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Central Ohio Urology Group, Gahanna, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - Lowcountry Urology Institute, Charleston, South Carolina
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Urology Associates of Nashville, Nashville, Tennessee
  - Urology of Virginia, Virginia Beach, Virginia
  - Spokane Urology, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Based on precedent, only IPD used in the results publication may be shared; however, the internal Dendreon team has not yet discussed this.

REFERENCES:
- See also: Dendreon Clinical Trial Summary Webpage — https://www.dendreon.com/science-and-services/provenge-prostate-cancer-immunotherapy/